CLINICAL TRIAL: NCT02477696
Title: A Randomized, Multicenter, Open-Label, Non-Inferiority, Phase III Study of Acalabrutinib (ACP-196) Versus Ibrutinib in Previously Treated Subjects With High Risk Chronic Lymphocytic Leukemia
Brief Title: Study of Acalabrutinib (ACP-196) Versus Ibrutinib in Previously Treated Participants With High Risk Chronic Lymphocytic Leukemia (CLL)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Acerta Pharma BV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ACE-CL-006; 2023-509347-27-00 (Registry Identifier: CTIS (EU)); 2014-005530-64 (EudraCT Number)
Record Dates: First submitted 2015-06-12; First posted 2015-06-23 (Estimated); Results first posted 2022-01-28 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — acalabrutinib; ibrutinib

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acalabrutinib (Experimental): Participants will receive oral acalabrutinib 100 mg twice daily (BID) until disease progression (PD), or unacceptable toxicity, or other reasons for discontinuation, whichever occurs first.
  Interventions: Drug: Acalabrutinib
- Ibrutinib (Active Comparator): Participants will receive oral ibrutinib 420 mg once daily (QD) until PD, or unacceptable toxicity, or other reasons for discontinuation, whichever occurrs first.
  Interventions: Drug: Ibrutinib

INTERVENTIONS:
Drug: Acalabrutinib — Participants will receive oral acalabrutinib as stated in arm description.
  Other Names: ACP-196
  Arms: Acalabrutinib
Drug: Ibrutinib — Participants will receive oral ibrutinib as stated in arm description.
  Arms: Ibrutinib

SUMMARY:
This study is designed to evaluate progression-free survival (PFS) endpoint for acalabrutinib versus (vs) ibrutinib in previously treated chronic lymphocytic leukemia.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥ 18 years of age.
* ECOG performance status of 0 to 2.
* Diagnosis of CLL.
* Must have ≥ 1 of the following high-risk prognostic factors:

  * Presence of 17p del by central laboratory.
  * Presence of 11q del by central laboratory.
* Active disease meeting ≥ 1 of the following IWCLL 2008 criteria for requiring treatment
* Must have received ≥ 1 prior therapies for CLL.
* Meet the following laboratory parameters:

  * Absolute neutrophil count (ANC) ≥ 750 cells/μL or ≥ 500 cells/μL in participants with documented bone marrow involvement, and independent of growth factor support 7 days before assessment.
  * Platelet count ≥ 30,000 cells/μL without transfusion support 7 days before assessment. Participants with transfusion-dependent thrombocytopenia are excluded.
  * Serum aspartate aminotransferase (AST)/serum glutamic oxaloacetic transaminase (SGOT) and alanine aminotransferase (ALT)/serum glutamic-pyruvic transaminase (SGPT) ≤ 3.0 x upper limit of normal (ULN).
  * Total bilirubin ≤ 1.5 x ULN.
  * Estimated creatinine clearance ≥ 30 mL/min.

Exclusion Criteria:

* Known CNS lymphoma or leukemia.
* Known prolymphocytic leukemia or history of, or currently suspected, Richter's syndrome.
* Uncontrolled autoimmune hemolytic anemia or idiopathic thrombocytopenia purpura.
* Prior exposure to ibrutinib or to a B-cell receptor (BCR) inhibitor or a B-cell lymphoma-2 (BCL-2) inhibitor.
* Received any chemotherapy, external beam radiation therapy, anticancer antibodies, or investigational drug within 30 days before first dose of study drug.
* Prior radio- or toxin-conjugated antibody therapy.
* Prior allogeneic stem cell or autologous transplant.
* Major surgery within 4 weeks before first dose of study drug.
* Prior malignancy, except for adequately treated lentigo maligna melanoma, non-melanomatous skin cancer, in situ cervical carcinoma or other malignancy treated with no evidence of active disease > 3 years before Screening and at low risk for recurrence.
* Significant cardiovascular disease within 6 months of screening.
* Known history of infection with human immunodeficiency virus (HIV).
* History of stroke or intracranial hemorrhage within 6 months before randomization.
* History of bleeding diathesis.
* Requires or receiving anticoagulation with warfarin or equivalent vitamin K antagonists within 7 days of first dose of study drug.
* Requires treatment with a strong cytochrome P450 3A (CYP3A) inhibitor/inducer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 533 (Actual)
Dates: Start 2015-07-28 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2028-01-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Acerta Clinical Trials, Study Director — 1-888-292-9613
Locations (118):
- United States (29):
  - Research Site, Phoenix, Arizona
  - Research Site, Anaheim, California
  - Research Site, Berkeley, California
  - Research Site, Duarte, California
  - Research Site, La Jolla, California
  - Research Site, Los Angeles, California
  - Research Site, Palo Alto, California
  - Research Site, Santa Rosa, California
  - Research Site, Jacksonville, Florida
  - Research Site, Tampa, Florida
  - Research Site, Athens, Georgia
  - Research Site, Harvey, Illinois
  - Research Site, Peoria, Illinois
  - Research Site, Wichita, Kansas
  - Research Site, Minneapolis, Minnesota
  - Research Site, Rochester, Minnesota
  - Research Site, Billings, Montana
  - Research Site, Hackensack, New Jersey
  - Research Site, Lake Success, New York
  - Research Site, New Hyde Park, New York
  - Research Site, New York, New York
  - Research Site, Durham, North Carolina
  - Research Site, Columbus, Ohio
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Houston, Texas
  - Research Site, Round Rock, Texas
  - Research Site, Charlottesville, Virginia
  - Research Site, Tacoma, Washington
  - Research Site, Northwest WA, Wisconsin
- Australia (6):
  - Research Site, Darlinghurst
  - Research Site, Frankston
  - Research Site, Melbourne
  - Research Site, St Leonards
  - Research Site, Waratah NSW
  - Research Site, Wollongong
- Belgium (5):
  - Research Site, Bruges
  - Research Site, Brussels
  - Research Site, Ghent
  - Research Site, Leuven
  - Research Site, Yvoir
- Denmark (2):
  - Research Site, Aalborg
  - Research Site, Indgang 27B
- France (6):
  - Research Site, Bobigny
  - Research Site, Créteil
  - Research Site, Pierre-Bénite
  - Research Site, Rennes
  - Research Site, Rouen
  - Research Site, Toulouse
- Germany (2):
  - Research Site, München
  - Research Site, Ulm
- Hungary (3):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Kaposvár
- Israel (6):
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Nahariya
  - Research Site, Petah Tikvah
  - Research Site, Tel Litwinsky
  - Research Site, Tiberias
- Italy (9):
  - Research Site, Bologna
  - Research Site, Cagliari
  - Research Site, Cona
  - Research Site, Florence
  - Research Site, Meldola
  - Research Site, Milan
  - Research Site, Modena
  - Research Site, Ravenna
  - Research Site, Rome
- Netherlands (13):
  - Research Site, Almere Stad
  - Research Site, Amsterdam
  - Research Site, Blaricum
  - Research Site, Breda
  - Research Site, Delft
  - Research Site, Dordrecht
  - Research Site, Geleen
  - Research Site, Groningen
  - Research Site, Haarlem
  - Research Site, Leiden
  - Research Site, Rotterdam
  - Research Site, Utrecht
  - Research Site, Zutphens
- New Zealand (3):
  - Research Site, Addington
  - Research Site, Auckland
  - Research Site, Tauranga
- Poland (9):
  - Research Site, Bydgoszcz
  - Research Site, Gdansk
  - Research Site, Gdynia
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Olsztyn
  - Research Site, Opole
  - Research Site, Słupsk
  - Research Site, Wroclaw
- Spain (5):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Majadahonda
  - Research Site, Murcia
  - Research Site, Santander
- Turkey (Türkiye) (5):
  - Research Site, Ankara
  - Research Site, Instabul
  - Research Site, Istanbul
  - Research Site, Izmir
  - Research Site, Kayseri
- United Kingdom (15):
  - Research Site, Birmingham
  - Research Site, Bournemouth
  - Research Site, Cambridge
  - Research Site, Cardiff
  - Research Site, Greater London
  - Research Site, Hull
  - Research Site, Leeds
  - Research Site, Leicester
  - Research Site, Liverpool
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Nottingham
  - Research Site, Plymouth
  - Research Site, Southampton
  - Research Site, Surrey

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Byrd JC, Hakre S, Ghia P. How well does acalabrutinib work and how safe is it to treat patients with chronic lymphocytic leukemia/small lymphocytic lymphoma who have had previous treatments? a plain language summary of 2 key studies. Future Oncol. 2025 Nov;21(26):3343-3357. doi: 10.1080/14796694.2025.2494976. Epub 2025 Jun 8. PMID 40485230
- [Derived] Alfaifi A, Bahashwan S, Alsaadi M, Ageel AH, Ahmed HH, Fatima K, Malhan H, Qadri I, Almehdar H. Advancements in B-Cell Non-Hodgkin's Lymphoma: From Signaling Pathways to Targeted Therapies. Adv Hematol. 2024 Nov 12;2024:5948170. doi: 10.1155/2024/5948170. eCollection 2024. PMID 39563886
- [Derived] Woyach JA, Jones D, Jurczak W, Robak T, Illes A, Kater AP, Ghia P, Byrd JC, Seymour JF, Long S, Mohamed N, Benrashid S, Lai TH, De Jesus G, Lai R, de Bruin G, Rule S, Munugalavadla V. Mutational profile in previously treated patients with chronic lymphocytic leukemia progression on acalabrutinib or ibrutinib. Blood. 2024 Sep 5;144(10):1061-1068. doi: 10.1182/blood.2023023659. PMID 38754046
- [Derived] Seymour JF, Byrd JC, Ghia P, Kater AP, Chanan-Khan A, Furman RR, O'Brien S, Brown JR, Munir T, Mato A, Stilgenbauer S, Bajwa N, Miranda P, Higgins K, John E, de Borja M, Jurczak W, Woyach JA. Detailed safety profile of acalabrutinib vs ibrutinib in previously treated chronic lymphocytic leukemia in the ELEVATE-RR trial. Blood. 2023 Aug 24;142(8):687-699. doi: 10.1182/blood.2022018818. PMID 37390310
- [Derived] Kipps TJ. Mining the Microenvironment for Therapeutic Targets in Chronic Lymphocytic Leukemia. Cancer J. 2021 Jul-Aug 01;27(4):306-313. doi: 10.1097/PPO.0000000000000536. PMID 34398557
- [Derived] Byrd JC, Hillmen P, Ghia P, Kater AP, Chanan-Khan A, Furman RR, O'Brien S, Yenerel MN, Illes A, Kay N, Garcia-Marco JA, Mato A, Pinilla-Ibarz J, Seymour JF, Lepretre S, Stilgenbauer S, Robak T, Rothbaum W, Izumi R, Hamdy A, Patel P, Higgins K, Sohoni S, Jurczak W. Acalabrutinib Versus Ibrutinib in Previously Treated Chronic Lymphocytic Leukemia: Results of the First Randomized Phase III Trial. J Clin Oncol. 2021 Nov 1;39(31):3441-3452. doi: 10.1200/JCO.21.01210. Epub 2021 Jul 26. PMID 34310172
- See also: Redacted CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=ACE-CL-006&attachmentIdentifier=939fcaa0-05d0-4eeb-901b-543dfc69a943&fileName=ace-cl-006-clinical-study-report_synopsis-redact.pdf&versionIdentifier=
- See also: Redacted CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=ACE-CL-006&attachmentIdentifier=48862a92-675d-444e-bdd0-df4a7b6c70b3&fileName=ace-cl-006-csp-v-amendment-5-global-redact.pdf&versionIdentifier=
- See also: Redacted SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=ACE-CL-006&attachmentIdentifier=62830b27-5baf-4d43-b70a-7b62304b80d0&fileName=ace-cl-006-SAP-redact.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 533 participants were randomized in this study of which 529 participants were treated (4 participants were randomized but not treated).
Groups:
- Acalabrutinib: Participants received oral acalabrutinib (ACP196) 100 mg twice daily (BID) until disease progression (PD), or unacceptable toxicity, or other reasons for discontinuation, whichever occurred first.
- Ibrutinib: Participants received oral ibrutinib 420 mg once daily (QD) until PD, or unacceptable toxicity, or other reasons for discontinuation, whichever occurred first.
Period: Overall Study
Arm/Group | Acalabrutinib | Ibrutinib
Started | 268 | 265
Treated | 265 | 264
Completed | 0 | 0
Not Completed | 268 | 265
Not completed — Death | 89 | 106
Not completed — Lost to Follow-up | 7 | 5
Not completed — Withdrawal by Subject | 37 | 34
Not completed — Physician Decision | 7 | 9
Not completed — Study terminated by sponsor | 103 | 99
Not completed — Other reasons including transition to commercial drug | 23 | 12
Not completed — Missing/Unknown | 2 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all participants randomized and were analyzed according to the arm to which they were randomly assigned.
Groups:
- Acalabrutinib: Participants received oral acalabrutinib (ACP196) 100 mg BID until PD, or unacceptable toxicity, or other reasons for discontinuation, whichever occurred first.
- Ibrutinib: Participants received oral ibrutinib 420 mg QD until PD, or unacceptable toxicity, or other reasons for discontinuation, whichever occurred first.
- Total: Total of all reporting groups
Arm/Group | Acalabrutinib | Ibrutinib | Total
Number analyzed (Participants) | 268 | 265 | 533
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Age (years) | 65.5 (9.3) | 65.3 (9.6) | 65.4 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Sex: Female | 83 | 71 | 154
  Sex: Male | 185 | 194 | 379
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 5 | 13
  Not Hispanic or Latino | 235 | 237 | 472
  Unknown or Not Reported | 25 | 23 | 48
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 8 | 13
  White | 257 | 245 | 502
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 10 | 15

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) Based on Independent Review Committee (IRC) Assessment
Description: The PFS is defined as the time from date of randomization to the date of first IRC-assessed PD or death due to any cause, whichever occurred first. PD (per International Workshop on Chronic Lymphocytic Leukemia [iwCLL] 2008 criteria): Lymphocytes >= 50% increase over baseline, or >= 50% increase in lymphadenopathy/hepatomegaly/splenomegaly, or >= 50% platelets or > 2 g/dL hemoglobin decreases from baseline secondary to chronic lymphocytic leukemia (CLL). The PFS is assessed using the Kaplan-Meier method.
Time Frame: Baseline (Days -28 to -1) through 55.2 months (maximum observed duration)
Population: ITT population included all participants randomized and were analyzed according to the arm to which they were randomly assigned.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Acalabrutinib | Ibrutinib
Number analyzed (Participants) | 268 | 265
Months | 38.4 [33.0 to 38.6] | 38.4 [33.0 to 41.6]
Statistical Analysis 1: Comparison: Acalabrutinib vs Ibrutinib; Test type: Non-Inferiority — Non-inferiority of acalabrutinib was demonstrated if the upper bound of the 2-sided 95% confidence interval (CI) of the hazard ratio was below 1.429; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.79 to 1.27] — Cox Proportional Hazards model stratified by 17p deletion status (yes versus no) and number of prior therapies (1-3 versus >=4)

2. Secondary Outcome: Number of Participants With Treatment-emergent Infections Grade >= 3
Description: Number of participants with treatment-emergent infections Grade >=3 are reported.
Time Frame: Day 1 through 83.5 months (maximum observed duration)
Population: Safety population included all participants who received at least one dose of study drug and were analyzed as treated.
Measure: Count of Participants; unit: Participants
Arm/Group | Acalabrutinib | Ibrutinib
Number analyzed (Participants) | 266 | 263
Participants | 98 | 101

3. Secondary Outcome: Number of Participants With Treatment-emergent Richter's Transformation
Description: Richter's transformation is defined as the occurrence of an aggressive lymphoma in participants with a previous or concomitant diagnosis of CLL. Richter's transformation was assessed by central pathology. Number of participants with treatment-emergent Richter's transformation are reported.
Time Frame: Day 1 through 83.5 months (maximum observed duration)
Population: Safety population included all participants who received at least one dose of study drug and were analyzed as treated.
Measure: Count of Participants; unit: Participants
Arm/Group | Acalabrutinib | Ibrutinib
Number analyzed (Participants) | 266 | 263
Participants | 13 | 14

4. Secondary Outcome: Number of Participants With Treatment-emergent Atrial Fibrillation
Description: Number of participants with treatment-emergent atrial fibrillation (including atrial flutter) are reported.
Time Frame: Day 1 through 83.5 months (maximum observed duration)
Population: Safety population included all participants who received at least one dose of study drug and were analyzed as treated.
Measure: Count of Participants; unit: Participants
Arm/Group | Acalabrutinib | Ibrutinib
Number analyzed (Participants) | 266 | 263
Participants | 32 | 49

5. Secondary Outcome: Overall Survival (OS)
Description: The OS is defined as the time from date of randomization to date of death due to any cause. The OS is assessed using the Kaplan-Meier method.
Time Frame: Baseline (Days -28 to -1) through 83.7 months (maximum observed duration)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Acalabrutinib | Ibrutinib
Number analyzed (Participants) | 268 | 265
Months | NA [NA to NA] — The median was not reached at the time of data cutoff. 95% CI was not calculable because an insufficient number of participants had event. | NA [65.0 to NA] — The median was not reached at the time of data cutoff. Upper limit of 95% CI was not calculable because an insufficient number of participants had event.

6. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. The TEAEs are defined as events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug.
Time Frame: Day 1 through 83.5 months (maximum observed duration)
Population: Safety population included all participants who received at least one dose of study drug and were analyzed as treated.
Measure: Count of Participants; unit: Participants
Arm/Group | Acalabrutinib | Ibrutinib
Number analyzed (Participants) | 266 | 263
Participants
  Any TEAEs | 262 | 259
  Any TESAEs | 161 | 177

7. Secondary Outcome: Number of Participants With Treatment-emergent Laboratory Abnormalities
Description: Number of participants with treatment-emergent laboratory abnormalities are reported. Laboratory abnormality is defined as any abnormal finding during analysis of hematology and serum chemistry.
Time Frame: Day 1 through 83.5 months (maximum observed duration)
Population: Safety population included all participants who received at least one dose of study drug and were analyzed as treated.
Measure: Count of Participants; unit: Participants
Arm/Group | Acalabrutinib | Ibrutinib
Number analyzed (Participants) | 266 | 263
Participants
  Absolute neutrophil count (decreased) | 124 | 135
  Haemoglobin (decreased) | 139 | 131
  Platelets (decreased) | 119 | 116
  Leukocytes (decreased) | 60 | 64
  Leukocytes (increased) | 68 | 84
  Absolute lymphocyte count (ALC) (decreased) | 66 | 65
  ALC (increased) | 71 | 72
  Alanine aminotransferase (increased) | 73 | 70
  Albumin (decreased) | 31 | 44
  Alkaline phosphatase (increased) | 66 | 60
  Aspartate aminotransferase (increased) | 42 | 58
  Bilirubin (increased) | 46 | 69
  Calcium (decreased) | 56 | 71
  Calcium (increased) | 15 | 11
  Creatinine (increased) | 164 | 168
  Glucose (decreased) | 5 | 13
  Glucose (increased) | 21 | 23
  Phosphate (decreased) | 93 | 74
  Potassium (decreased) | 27 | 40
  Potassium (increased) | 62 | 52
  Sodium (decreased) | 26 | 37
  Sodium (increased) | 70 | 46
  Urate (increased) | 70 | 96

8. Secondary Outcome: Number of Participants With Abnormal Vital Signs Reported as TEAEs
Description: Number of participants with abnormal vital signs reported as TEAEs are reported. Abnormal vital signs are defined as any abnormal finding in the vital sign parameters (body temperature, blood pressure, heart rate, and respiratory rate).
Time Frame: Day 1 through 83.5 months (maximum observed duration)
Population: Safety population included all participants who received at least one dose of study drug and were analyzed as treated.
Measure: Count of Participants; unit: Participants
Arm/Group | Acalabrutinib | Ibrutinib
Number analyzed (Participants) | 266 | 263
Participants
  Abnormal loss of weight | 0 | 1
  Blood pressure fluctuation | 0 | 1
  Blood pressure increased | 2 | 3
  Blood pressure decreased | 1 | 0
  Blood pressure systolic increased | 0 | 1
  Body temperature decreased | 1 | 0
  Body temperature increased | 0 | 1
  Bradycardia | 3 | 1
  Breath sounds abnormal | 0 | 1
  Cardiac murmur | 1 | 2
  Dyspnoea | 40 | 27
  Dyspnoea exertional | 2 | 5
  Heart rate increased | 0 | 1
  Heart rate irregular | 1 | 0
  Hypertension | 26 | 70
  Hypotension | 15 | 7
  Hyperpyrexia | 1 | 0
  Orthostatic hypotension | 2 | 1
  Palpitations | 12 | 15
  Pyrexia | 66 | 55
  Tachycardia | 7 | 7
  Weight decreased | 29 | 23
  Weight increased | 13 | 10
  White coat hypertension | 0 | 1

9. Secondary Outcome: Percentage of Participants With Lymphocytosis
Description: Percentage of participants with at least one occurrence of treatment-related lymphocytosis defined as an elevation in ALC of >= 50% compared with baseline and a postbaseline assessment of > 5000/μL in the peripheral blood are reported.
Time Frame: Day 1 through 83.5 months (maximum observed duration)
Population: Safety population included all participants who received at least one dose of study drug and were analyzed as treated.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Acalabrutinib | Ibrutinib
Number analyzed (Participants) | 266 | 263
Percentage of participants | 72.5 [66.7 to 77.7] | 74.3 [68.6 to 79.5]

10. Secondary Outcome: Number of Participants With Electrocardiogram (ECG) Abnormality at Baseline
Description: Number of participants with ECG abnormality at baseline are reported.
Time Frame: Baseline (Days -28 to -1)
Population: Safety population included all participants who received at least one dose of study drug and were analyzed as treated.
Measure: Count of Participants; unit: Participants
Arm/Group | Acalabrutinib | Ibrutinib
Number analyzed (Participants) | 266 | 263
Participants
  Abnormal, not clinically significant | 86 | 98
  Abnormal, clinically significant | 4 | 1

11. Secondary Outcome: Number of Participants With Shift From Baseline to Worst (Grade 3 and 4) Postbaseline in Eastern Cooperative Oncology Group (ECOG) Performance Status
Description: The ECOG performance status assessed participant's performance status on 5 point scale: 0=Fully active/able to carry on all pre-disease activities without restriction; 1=restricted in physically strenuous activity, ambulatory/able to carry out light or sedentary work; 2=ambulatory (>50% of waking hours), capable of all self-care, unable to carry out any work activities; 3=capable of only limited self care, confined to bed/chair >50% of waking hrs; 4=completely disabled, cannot carry on any self care, totally confined to bed/chair; 5=death. Number of participants with shift from baseline (Days -28 to -1) to worst Grade 3 and 4 in ECOG performance status are reported.
Time Frame: Baseline (Days -28 to -1) through 83.5 months (maximum observed duration)
Population: Safety population included all participants who received at least one dose of study drug and were analyzed as treated. Here, "number of participants analyzed" (N) signified those participants who had a baseline value and at least 1 postbaseline value of ECOG performance status score during the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Acalabrutinib | Ibrutinib
Number analyzed (Participants) | 259 | 253
Participants
  Baseline=0; Postbaseline=3 | 0 | 1
  Baseline=1; Postbaseline=3 | 3 | 5
  Baseline=2; Postbaseline=3 | 4 | 1
  Baseline=0; Postbaseline=4 | 0 | 0
  Baseline=1; Postbaseline=4 | 0 | 0
  Baseline=2; Postbaseline=4 | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 through 83.5 months (maximum observed duration).
Description: The AE/SAE data are reported for safety population. Safety population included all participants who received at least one dose of study drug and were analyzed as treated.
Arm/Group | Acalabrutinib | Ibrutinib
All-Cause Mortality (participants affected / at risk) | 89/266 | 106/263
Serious Adverse Events (participants affected / at risk) | 161/266 | 177/263
Other Adverse Events (participants affected / at risk) | 251/266 | 251/263
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acalabrutinib (N=266) | Ibrutinib (N=263)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 1 (2)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 2 (2)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Aspergillus infection (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1)
Bacterial sepsis (Infections and infestations) | 0 (0) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 6 (6) | 3 (3)
Biliary sepsis (Infections and infestations) | 0 (0) | 1 (1)
Blister infected (Infections and infestations) | 1 (2) | 0 (0)
Bone abscess (Infections and infestations) | 0 (0) | 1 (1)
Brain abscess (Infections and infestations) | 2 (2) | 0 (0)
Bronchitis (Infections and infestations) | 4 (4) | 2 (2)
Bronchopulmonary aspergillosis (Infections and infestations) | 2 (2) | 1 (1)
COVID-19 (Infections and infestations) | 15 (17) | 14 (14)
COVID-19 pneumonia (Infections and infestations) | 2 (2) | 5 (6)
Campylobacter infection (Infections and infestations) | 0 (0) | 1 (2)
Cellulitis (Infections and infestations) | 3 (3) | 4 (5)
Thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cellulitis staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Cerebral aspergillosis (Infections and infestations) | 1 (1) | 1 (1)
Chronic sinusitis (Infections and infestations) | 1 (1) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 2 (2) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 2 (3) | 1 (1)
Coccidioidomycosis (Infections and infestations) | 0 (0) | 1 (1)
Cryptococcosis (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Dermatitis infected (Infections and infestations) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 3 (4) | 1 (1)
Diarrhoea infectious (Infections and infestations) | 1 (1) | 0 (0)
Encephalitis viral (Infections and infestations) | 0 (0) | 1 (1)
Epstein-barr virus infection reactivation (Infections and infestations) | 0 (0) | 1 (1)
Escherichia pyelonephritis (Infections and infestations) | 0 (0) | 1 (2)
Escherichia sepsis (Infections and infestations) | 2 (2) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 3 (3) | 2 (2)
Fungal abscess central nervous system (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 2 (2)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0)
Groin abscess (Infections and infestations) | 1 (1) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Haematoma infection (Infections and infestations) | 0 (0) | 1 (1)
Haemophilus infection (Infections and infestations) | 1 (1) | 1 (1)
Hepatitis e (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 2 (2)
Herpes zoster meningoencephalitis (Infections and infestations) | 1 (1) | 0 (0)
Hydrocele male infected (Infections and infestations) | 0 (0) | 1 (1)
Infected bite (Infections and infestations) | 0 (0) | 1 (2)
Infected skin ulcer (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 2 (2)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 8 (9) | 16 (17)
Infective exacerbation of bronchiectasis (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 3 (3) | 3 (3)
Klebsiella sepsis (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (2) | 4 (7)
Lymphadenitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Meningitis (Infections and infestations) | 0 (0) | 1 (1)
Metapneumovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Necrotising ulcerative gingivostomatitis (Infections and infestations) | 1 (1) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 2 (2) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Nocardiosis (Infections and infestations) | 0 (0) | 1 (1)
Norovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Oral fungal infection (Infections and infestations) | 1 (1) | 0 (0)
Orchitis (Infections and infestations) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 1 (1) | 0 (0)
Parainfluenzae virus infection (Infections and infestations) | 0 (0) | 2 (2)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 1 (1)
Picornavirus infection (Infections and infestations) | 1 (1) | 0 (0)
Atrioventricular block (Cardiac disorders) | 0 (0) | 1 (1)
Pneumococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 5 (5) | 0 (0)
Pneumonia (Infections and infestations) | 33 (56) | 30 (45)
Pneumonia acinetobacter (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 2 (2) | 1 (1)
Pneumonia haemophilus (Infections and infestations) | 1 (1) | 2 (2)
Pneumonia influenzal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia klebsiella (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia mycoplasmal (Infections and infestations) | 1 (1) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 1 (1) | 1 (1)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia pseudomonal (Infections and infestations) | 5 (6) | 0 (0)
Pneumonia staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia streptococcal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0)
Post procedural cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1) | 1 (1)
Pseudomonal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary nocardiosis (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Bradyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Rhinovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Salmonella sepsis (Infections and infestations) | 0 (0) | 1 (2)
Sepsis (Infections and infestations) | 5 (5) | 7 (8)
Septic shock (Infections and infestations) | 2 (2) | 2 (2)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 0 (0) | 2 (2)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Stenotrophomonas infection (Infections and infestations) | 1 (1) | 0 (0)
Systemic infection (Infections and infestations) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 15 (15) | 13 (16)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 2 (2)
Urinary tract candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3) | 7 (9)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 1 (2)
Urinary tract infection enterococcal (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection pseudomonal (Infections and infestations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 2 (3) | 1 (1)
Varicella zoster virus infection (Infections and infestations) | 0 (0) | 2 (2)
Viral pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Bundle branch block (Cardiac disorders) | 0 (0) | 1 (1)
Wound infection bacterial (Infections and infestations) | 1 (2) | 0 (0)
Wound infection staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 2 (2) | 3 (3)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Splenic rupture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Subdural haematoma (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Cardiac asthma (Cardiac disorders) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 0 (0)
Blood magnesium decreased (Investigations) | 0 (0) | 1 (1)
Clostridium test positive (Investigations) | 1 (1) | 0 (0)
Glomerular filtration rate decreased (Investigations) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Cardiac failure (Cardiac disorders) | 4 (6) | 6 (6)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (2) | 3 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hypophagia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint instability (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (5)
Benign mesenteric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Burkitt's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Endometrial adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Leukaemic infiltration pulmonary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (5) | 2 (2)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 2 (2)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Polycythaemia vera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 6 (6)
Myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0)
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Squamous cell carcinoma of the parotid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma of the vulva (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Thymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 2 (2)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 3 (3) | 2 (2)
Cerebrovascular disorder (Nervous system disorders) | 0 (0) | 1 (1)
Demyelinating polyneuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Facial paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Guillain-barre syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 2 (2) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 4 (4)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Language disorder (Nervous system disorders) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1)
Multifocal motor neuropathy (Nervous system disorders) | 0 (0) | 1 (4)
Muscle spasticity (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Partial seizures (Nervous system disorders) | 0 (0) | 1 (1)
Post herpetic neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (2)
Pericardial effusion (Cardiac disorders) | 2 (2) | 2 (2)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 3 (4) | 4 (4)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 2 (2)
Confusional state (Psychiatric disorders) | 1 (2) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (3) | 6 (6)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 2 (2)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 2 (2)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 2 (2)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Oedema genital (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (2)
Vulvar dysplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 3 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Mediastinal haematoma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 5 (7)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary granuloma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary haematoma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Arteriovenous malformation (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Tonsillar disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Sudden hearing loss (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Aortic disorder (Vascular disorders) | 0 (0) | 1 (1)
Aortic dissection (Vascular disorders) | 0 (0) | 1 (1)
Circulatory collapse (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 1 (1)
Embolism venous (Vascular disorders) | 1 (1) | 0 (0)
Haemorrhagic infarction (Vascular disorders) | 1 (1) | 0 (0)
Hypercalcaemia of malignancy (Endocrine disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (2) | 1 (1)
Superficial vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1)
Vasculitis (Vascular disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Dacryoadenitis acquired (Eye disorders) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 4 (4)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal wall haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (5) | 6 (6)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 3 (4)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Erosive oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 3 (3)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Mallory-weiss syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pharyngo-oesophageal diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pneumatosis intestinalis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (2)
Sigmoid mesocolon hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Splenic artery aneurysm (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Volvulus (Gastrointestinal disorders) | 0 (0) | 1 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 2 (2)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (2) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 0 (0) | 2 (2)
Malaise (General disorders) | 0 (0) | 1 (1)
Mass (General disorders) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
Pyrexia (General disorders) | 11 (11) | 6 (6)
Soft tissue inflammation (General disorders) | 1 (1) | 0 (0)
Tissue infiltration (General disorders) | 0 (0) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 2 (2) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Amyloidosis (Immune system disorders) | 0 (0) | 1 (1)
Food allergy (Immune system disorders) | 0 (0) | 1 (1)
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acalabrutinib (N=266) | Ibrutinib (N=263)
Hypogammaglobulinaemia (Immune system disorders) | 13 (16) | 15 (17)
Thrombocytopenia (Blood and lymphatic system disorders) | 38 (70) | 36 (60)
Bronchitis (Infections and infestations) | 35 (58) | 23 (28)
COVID-19 (Infections and infestations) | 29 (34) | 24 (28)
Conjunctivitis (Infections and infestations) | 12 (13) | 15 (19)
Herpes zoster (Infections and infestations) | 24 (25) | 16 (19)
Atrial fibrillation (Cardiac disorders) | 26 (33) | 42 (48)
Influenza (Infections and infestations) | 11 (14) | 15 (18)
Lower respiratory tract infection (Infections and infestations) | 9 (17) | 19 (37)
Nasopharyngitis (Infections and infestations) | 30 (42) | 28 (35)
Oral herpes (Infections and infestations) | 18 (22) | 17 (18)
Pneumonia (Infections and infestations) | 33 (47) | 32 (40)
Respiratory tract infection (Infections and infestations) | 12 (12) | 14 (21)
Sinusitis (Infections and infestations) | 26 (36) | 22 (35)
Anaemia (Blood and lymphatic system disorders) | 53 (95) | 48 (86)
Upper respiratory tract infection (Infections and infestations) | 73 (122) | 65 (106)
Urinary tract infection (Infections and infestations) | 24 (47) | 38 (76)
Contusion (Injury, poisoning and procedural complications) | 31 (43) | 47 (66)
Fall (Injury, poisoning and procedural complications) | 14 (20) | 10 (14)
Weight decreased (Investigations) | 29 (35) | 23 (30)
Decreased appetite (Metabolism and nutrition disorders) | 19 (26) | 26 (33)
Hyperuricaemia (Metabolism and nutrition disorders) | 17 (17) | 19 (23)
Hypokalaemia (Metabolism and nutrition disorders) | 13 (13) | 25 (32)
Arthralgia (Musculoskeletal and connective tissue disorders) | 55 (84) | 70 (120)
Back pain (Musculoskeletal and connective tissue disorders) | 27 (32) | 40 (44)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 16 (19) | 41 (66)
Myalgia (Musculoskeletal and connective tissue disorders) | 25 (37) | 24 (37)
Neck pain (Musculoskeletal and connective tissue disorders) | 14 (14) | 6 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 23 (31) | 28 (45)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 14 (19) | 13 (17)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 14 (21) | 9 (11)
Dizziness (Nervous system disorders) | 30 (48) | 27 (41)
Palpitations (Cardiac disorders) | 11 (17) | 15 (17)
Headache (Nervous system disorders) | 92 (164) | 56 (100)
Paraesthesia (Nervous system disorders) | 14 (20) | 11 (16)
Insomnia (Psychiatric disorders) | 28 (31) | 13 (14)
Cough (Respiratory, thoracic and mediastinal disorders) | 79 (118) | 60 (93)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 37 (47) | 26 (35)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 22 (30) | 29 (47)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 18 (26) | 16 (21)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 22 (28) | 20 (23)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 20 (26) | 14 (15)
Ecchymosis (Skin and subcutaneous tissue disorders) | 14 (20) | 11 (13)
Onychoclasis (Skin and subcutaneous tissue disorders) | 2 (2) | 18 (20)
Petechiae (Skin and subcutaneous tissue disorders) | 12 (15) | 24 (26)
Pruritus (Skin and subcutaneous tissue disorders) | 16 (17) | 12 (14)
Rash (Skin and subcutaneous tissue disorders) | 27 (37) | 35 (50)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 12 (18) | 15 (18)
Haematoma (Vascular disorders) | 24 (47) | 20 (28)
Hypertension (Vascular disorders) | 26 (41) | 70 (118)
Hypotension (Vascular disorders) | 14 (17) | 7 (8)
Cataract (Eye disorders) | 12 (18) | 17 (23)
Abdominal pain (Gastrointestinal disorders) | 21 (24) | 21 (38)
Abdominal pain upper (Gastrointestinal disorders) | 17 (25) | 18 (21)
Constipation (Gastrointestinal disorders) | 33 (47) | 39 (48)
Diarrhoea (Gastrointestinal disorders) | 93 (180) | 122 (236)
Dyspepsia (Gastrointestinal disorders) | 12 (12) | 35 (39)
Nausea (Gastrointestinal disorders) | 49 (87) | 50 (63)
Increased tendency to bruise (Blood and lymphatic system disorders) | 5 (6) | 14 (17)
Stomatitis (Gastrointestinal disorders) | 9 (9) | 23 (28)
Toothache (Gastrointestinal disorders) | 6 (9) | 14 (17)
Vomiting (Gastrointestinal disorders) | 29 (38) | 36 (46)
Asthenia (General disorders) | 24 (37) | 27 (30)
Chills (General disorders) | 10 (12) | 17 (18)
Fatigue (General disorders) | 62 (89) | 48 (76)
Influenza like illness (General disorders) | 16 (23) | 16 (22)
Oedema peripheral (General disorders) | 33 (52) | 42 (58)
Neutropenia (Blood and lymphatic system disorders) | 56 (151) | 65 (156)
Pyrexia (General disorders) | 61 (97) | 50 (83)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.

DOCUMENTS (2):
  • Study Protocol (2020-10-21): https://cdn.clinicaltrials.gov/large-docs/96/NCT02477696/Prot_002.pdf
  • Statistical Analysis Plan (2020-10-23): https://cdn.clinicaltrials.gov/large-docs/96/NCT02477696/SAP_003.pdf